CLINICAL TRIAL: NCT04250129
Title: IS SENTINEL LYMPH NODE BIOPSY WITH RADIOTHERAPY ALONE WITHOUT AXILLARY LYMPH NODE DISSECTION SAFE FOLLOWING NEOADJUVANT CHEMOTHERAPY IN INITIALLY CLINICALLY AXILLA POSITIVE PATIENTS: NEOSENTITURK-TRIAL/MF-18-03
Brief Title: SENTINEL LYMPH NODE BIOPSY AFTER NEOADJUVANT CHEMOTHERAPY
Acronym: NEOSENTITURK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federation of Breast Diseases Societies (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-03
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Sentinel Lymph Node
Keywords: sentinel lymph node biopsy, Neoadjuvan chemotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SLNB (-)&level 1-3 RT: SLNB (-)&level 1-3 RT
- SLNB (+)&level 1-3 RT: SLNB (+)&level 1-3 RT
- SLNB(+)&ALND&level 3 RT (+/-level 1-2): SLNB(+)&ALND&level 3 RT (+/-level 1-2)

SUMMARY:
Omitting axilary lymph node dissection (ALND) following SLNB with residual cancer in patients with locally advanced disease after neoadjuvan chemotherapy (NAC) is still controversial. In this study, the investigators evaluated factors affecting local recurrence and outcome in patients with locally advanced breast cancer (LABC), who underwent sentinel lymph node (SLN) with or without ALND after NAC.

DETAILED DESCRIPTION:
All patients with clinically positive axilla will undergo neoadjuvant chemotherapy. Axillary fine needle aspiration biopsy or Trucut biopsy is mandatory.

All patients with clinically node negativity (physical exam, USG, and/or MRI, PET-CT) after Neoadjuvant Chemotherapy (NAC) will be considered for SLNB with any technique (blue dye alone, radionuclide alone or both combined) and any breast surgery (mastectomy or breast conservation). PET-CT and MRI are not mandatory. PE and USG and/or MRI are preferred. At least, 2 sentinel lymph nodes will be obtained. Intraoperative evaluation of SLNs is recommended.

All patients with clinally-negative axilla and underwent SLNB will be included into the study:

1. SLNB (-) & RT
2. SLNB (+) & RT
3. SLNB (+) & ALND & RT Radiotherapy details will be announced as supplementary

ELIGIBILITY:
Inclusion Criteria:

T0-4, N1-3, M0

Exclusion Criteria:

Inflammatory breast cancer, pregnant patients Patients with metastatic disease

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with clinically positive axilla will undergo neoadjuvant chemotherapy. All patients with clinically node negativity (physical exam, USG, and/or MRI, PET-CT) after Neoadjuvant Chemotherapy (NAC) will be considered for SLNB with any technique (blue dye alone, radionuclide alone or both combined) and any breast surgery (mastectomy or breast conservation). PET-CT and MRI are not mandatory. PE and USG and/or MRI are preferred. At least, 2 sentinel lymph nodes will be obtained. Intraoperative evaluation of SLNs is recomended.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Local recurrence free survival | January 2023
  Breast and axillary recurrence rates

SECONDARY OUTCOMES:
Disease free survival | January 2023
  Local recurrence and distant metastasis rates
Overall survival | January 2023
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Cabioglu, Prof, Principal Investigator — Istanbul University; Hasan Karanlik, Study Director — Istanbul University Institute of Oncology; Guldeniz Karadeniz Cakmak, Study Chair — Bulent Ecevit University Faculty of Medicine
Locations (3):
- Turkey (Türkiye) (3):
  - Istanbul University Institute of Oncology, Istanbul
  - Istanbul University Istanbul Faculty of Medicine, Istanbul
  - Bulent Ecevit University Faculty of Medicine, Zonguldak